CLINICAL TRIAL: NCT06466317
Title: Response of Metabolic Syndrome Components to Adding Honey Consumption to Free Walking Exercise in Children
Brief Title: Is There Effect of Adding Honey Intake to Free Walking in Metabolic Syndrome Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Hagar Ahmed El-Hadidy, Lecturer of Physical Therapy for Internal Medicine and Geriatrics, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T -PED-06/2024- 545
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey intake with walking exercise (Experimental): 20 Children with metabolic syndrome will receive free walking continuous exercise (thirty minutes daily in nearby sport club in the presence of their parents and walking will supervised by authors via Videoconferencing Imo Program) and this group also will healthy diet guidelines in addition to consuming natural honey (2ml/kg honey will be taken.. This dose will be divided into two halves, the first half will be taken at 7 am and the other half will be taken at 7 pm for 12 weeks)
  Interventions: Behavioral: Honey intake with walking exercise
- walking exercise (Active Comparator): 20 Children with metabolic syndrome will receive free walking continuous exercise (thirty minutes daily in nearby sport club in the presence of their parents and walking will supervised by authors via Videoconferencing Imo Program) and this group also will healthy diet guidelines for 12 weeks
  Interventions: Behavioral: Walking exercise

INTERVENTIONS:
Behavioral: Honey intake with walking exercise — 20 Children with metabolic syndrome will receive free walking continuous exercise (thirty minutes daily in nearby sport club in the presence of their parents and walking will supervised by authors via Videoconferencing Imo Program) and this group also will healthy diet guidelines in addition to consuming natural honey (2ml/kg honey will be taken.. This dose will be divided into two halves, the first half will be taken at 7 am and the other half will be taken at 7 pm for 12 weeks)
  Arms: Honey intake with walking exercise
Behavioral: Walking exercise — 20 Children with metabolic syndrome will receive free walking continuous exercise (thirty minutes daily in nearby sport club in the presence of their parents and walking will supervised by authors via Videoconferencing Imo Program) and this group also will healthy diet guidelines for 12 weeks)
  Arms: walking exercise

SUMMARY:
Metabolic Syndrome is common in Children and complementary therapies are important in its treatment such exercise and functional food intake including honey.

DETAILED DESCRIPTION:
Forty Children with metabolic syndrome will Assigned to group of free walking continuous exercise (thirty minutes daily in nearby sport club in the presence of their parents and walking was supervised by authors via Videoconferencing Imo Program) and this group also will receive healthy dietary guidelines in addition to consuming natural honey for 12 weeks.. The other group that will contain 20 patients will take only free walking exercise and healthy diet guidelines for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 40 metabolic syndrome children

Exclusion Criteria:

* respiratory, cardiac , renal , liver problems

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
high density lipoprotein | it will be assessed after 12 weeks
  it is a component of lipid profile

SECONDARY OUTCOMES:
triglycrides | it will be assessed after 12 weeks
  it is a component of lipid profile
body mass index | it will be assessed after 12 weeks
  it will be measured in morning with empty stomach and badder
waist circumference | it will be assessed after 12 weeks
  it will be measured by a tape at the level of umblicus
systolic blood pressure | it will be assessed after 12 weeks
  it will be measured by manual sphygomamnaometer
diastolic blood pressure | it will be assessed after 12 weeks
  it will be measured by manual sphygomamnaometer
fasting blood glucose | it will be assessed after 12 weeks
  it will be measured at morning

CONTACTS AND LOCATIONS:
Overall Officials: hagar el-hadidy, lecturer, Principal Investigator — Faculty of Physical Therapy, Ahram Canadian University (ACU), Giza, Egypt
Locations (1):
- Ahram canadian university, Giza, Egypt